CLINICAL TRIAL: NCT03133000
Title: Mini- or Less-Open Sublay Operation (MILOS) - a New Minimally Invasive Technique for the Extraperitoneal Repair of Incisional Hernias
Brief Title: Mini- or Less-Open Sublay Operation (MILOS) of Incisional Hernias
Status: Completed | Type: Observational
Sponsor: Gross Sand Hospital (Other)
Responsible Party: Principal Investigator, Wolfgang Reinpold, Director of the Department of Surgery and Hernia Center Gross Sand Hospital, Gross Sand Hospital
Other Study IDs: MILOS-Incisional-Hernia-2010
Record Dates: First submitted 2017-04-17; First posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Incisional Hernia
Keywords: Recurrent abdominal wall hernia; Incisional hernia
MeSH Terms: conditions — Incisional Hernia; Hernia, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective non-randomized observational register study of all elective symptomatic incisional hernias operated on in the Hernia Center of Reference of Gross Sand Hospital using the novel endoscopic assisted Mini- or Less-Open Sublay technique. The data of all patients were prospectively documented in the German Hernia Registry "Herniamed". The novel MILOS-technique allows the minimal invasive implantation of large extraperitoneal meshes for the treatment of primary and secondary incisional hernias.

DETAILED DESCRIPTION:
Prospective non-randomized observational register study of all elective symptomatic incisional hernias operated on in the Reference Hernia Center of Gross Sand Hospital between 1 January 2010 and 30 September 2015 using the novel endoscopic assisted Mini- or Less-Open Sublay technique. The novel MILOS-technique allows the minimal invasive implantation of large extraperitoneal meshes for the treatment of primary and secondary incisional hernias.The data of all patients were prospectively documented in the German Hernia Registry "Herniamed". Data privacy protection was strictly implemented according to German federal law. All patients were informed in detail about the new surgical technique, other treatment options, prospective register study with one year questionnaire follow-up, data documentation. All patients gave written consent.

A propensity score matching of all patients of the MILOS-cohort of Gross Sand Hospital with patients with comparable incisional hernias who were operated on using the laparoscopic intraperitoneal onlay mesh (IPOM) technique or open sublay technique in other institutions participating in the German Hernia Database "Herniated" was performed.

ELIGIBILITY:
Inclusion Criteria:

* All patients with symptomatic elective primary or secondary incisional hernias:
* Median incisional hernias
* Lateral incisional hernias

Exclusion Criteria:

* Emergencies
* Very large incisional hernias that required incisions larger than 12 cm

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with symptomatic elective incisional hernias who were referred to Gross Sand Hernia Center of Reference
Sampling Method: Non-Probability Sample
Enrollment: 615 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Recurrence after incisional hernia repair as assess by clinical examination at one year | one year follow-up
  Data collected in German National Hernia Registry (Herniamed)
Chronic pain after incisional hernia repair as reported by questionnaire and follow up examination at one year | one year follow-up
  Data collected in German National Hernia Registry (Herniamed)
Perioperative complications after incisional hernia repair | one year follow-up
  Data collected in German National Hernia Registry (Herniamed)
Reoperation after incisional hernia repair | one year follow-up
  Data collected in German National Hernia Registry (Herniamed)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Reinpold, Dr. MD, Study Director — Department of Surgery and Hernia Center Gross Sand Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reinpold W, Berger C, Adolf D, Kockerling F. Mini- or less-open sublay (E/MILOS) operation vs open sublay and laparoscopic IPOM repair for the treatment of incisional hernias: a registry-based propensity score matched analysis of the 5-year results. Hernia. 2024 Feb;28(1):179-190. doi: 10.1007/s10029-023-02847-3. Epub 2023 Aug 21. PMID 37603090
- [Derived] Reinpold W, Schroder M, Berger C, Nehls J, Schroder A, Hukauf M, Kockerling F, Bittner R. Mini- or Less-open Sublay Operation (MILOS): A New Minimally Invasive Technique for the Extraperitoneal Mesh Repair of Incisional Hernias. Ann Surg. 2019 Apr;269(4):748-755. doi: 10.1097/SLA.0000000000002661. PMID 29342018
- See also: Related Info — https://milos-hernia-repair.com/de/das-minimal-invasive-milos-verfahren